CLINICAL TRIAL: NCT04481763
Title: A Study of the Efficacy and Safety of Camrelizumab Plus Radiotherapy for Patients With Early Triple-Negative Breast
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCL2020
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab + radiotherapy (Other): This is a open-labeled, single-arm, Investigator-initiated clinical trial ,Compared with historical data
  Interventions: Drug: Camrelizumab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is 200 mg iv. administered every 2 weeks for 3 cycles with radiotherapy ( 50gy, 25 times for 5weeks)
Radiation: radiotherapy — radiotherapy

SUMMARY:
This is a open-labeled, single-arm, Investigator-initiated clinical trial of camrelizumab (an anti-PD-1 antibody) in combination with radiotherapy in patients with early triple-negative breast cancer. We will enroll 60 subjects. This study aims to evaluate the efficacy and safety of camrelizumab combined with radiotherapy in the treatment of early TNBC。

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, and exploratory clinical study, taking the Cancer Hospital of Jiangxi province as the lead unit, combined with breast cancer diagnosis and treatment norms, multi-center collaborative research to explore the iDFS of radiotherapy combined with carilizumab for triple-negative breast cancer of different subtypes and provide optimal personalized treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. female participants aged ≥ 18 years and < 75 years
2. Participants with a histological or cytological diagnosis of TNBC breast cancer , defined by ER <1%, PR <1% and HER2 negative on IHC and/or non-amplified by ISH by local lab testing
3. Gene detection for Subtypes of TNBC、PD-L1expression and TMB expression
4. Breast-conserving therapy is planned after mastectomy 1) largest focus must measure of Primary tumor ≥ 5cm，Tumor invades breast skin and chest wall 2) Axillary lymph node metastasis≥4 3) 1 -3 lymph node metastases in stage T1-2 4) Simple mastectomy combined with axillary lymphadenectomy in stage T1-2 (axillary lymph nodes are positive, and subsequent axillary dissection is not considered)
5. Adequate Organ Function as defined in the table below:

   Absolute neutrophil count (ANC) ≥ 1500/uL Platelet count ≥ 100,000/uL Hemoglobin ≥5.6mmol/L（9.0g/dL) serum albumin ≥2.8g/dL Serum creatinine ≤ ≤1.5mg/d or creatinine clearance ≥ 50mL/min Serum Total Bilirubin ≤ 1.5 X ULN AST&ALT≤2.5ULN
6. 12 lead ECG: friderica corrected QT interval (QTCF) < 470 Ms
7. Women of childbearing potential must have a negative urine or serum pregnancy test within 28 day prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 90 days after the last dose of study medication.
8. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Known additional malignancy that is progressing or has required active treatment .

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
2. Patients with evident metastatic lesions at the time of diagnosis
3. Has received prior therapy with an anti-PD-1, anti-PD-L1.History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
4. There are any active autoimmune diseases or a medical history of autoimmune (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid function Decreased. Subjects with vitiligo or adults who have had childhood asthma but have fully relieved without any intervention may be included. However, subjects who require bronchodilators for medical intervention cannot be included.)
5. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Ascites or pleural effusion with clinical symptoms, requiring therapeutic puncture or drainage
7. Cardiac clinical symptoms or diseases that are not well controlled, such as: a. Heart Failure NYHA > Class Ⅱ, b. unstable angina, c. myocardial infarction within 1 year; d. Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.
8. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), with obvious bleeding tendency or undergoing thrombolytic or anticoagulant treatment
9. History of clear tendency of gastrointestinal hemorrhage and active bleeding in unresected tumor within 3 months prior to the start of study treatment. for example, esophageal varices, gastric and duodenal active ulcer, ulcerative colitis, portal hypertension ; Or other conditions that may cause gastrointestinal bleeding and perforation determined by the researchers;
10. Previous or current serious bleeding (bleeding > 30ml in 3 months), hemoptysis (fresh blood > 5ml in 4 weeks) or thromboembolism within 12 months (including stroke events and / or transient ischemic attacks);
11. The patient has active infection during screening period, or unexplained fever (≥38.5 °C) before first administration ( According to the judgment of the researcher, the fever caused by the tumor can be included in the group);
12. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 4 weeks prior to the start of study treatment;
13. Has a history of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan.
14. Subjects with congenital or acquired immunodeficiency (such as HIV-infected), or active hepatitis (hepatitis B reference: HBsAg-positive, HBV DNA ≥ 2000 IU/ml or copy number ≥ 104/ml; hepatitis C reference: HCV antibody-positive.)
15. Patients who are participating in other clinical trials or less than 1 month from the end of the previous clinical study; Patients may receive other systemic anti-tumor treatment during the study period
16. Receive live vaccine within 4 weeks before or during the study period;
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. According to the investigator's assessment, there are other factors that may lead to the termination of the study, such as other serious diseases (including mental illness) requiring combined treatment. Any other condition and social/psychological problems, etc., the investigator judged that the patient was not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) | 3 years
  time from surgery to the first documented occurrence of an event, defined as: Ipsilateral invasive breast tumor recurrence, Ipsilateral local-regional invasive breast cancer recurrence, Distant recurrence, Contralateral invasive breast cancer, Death from any cause
Invasive disease-free survival (iDFS) | 5years
  time from surgery to the first documented occurrence of an event, defined as: Ipsilateral invasive breast tumor recurrence, Ipsilateral local-regional invasive breast cancer recurrence, Distant recurrence, Contralateral invasive breast cancer, Death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 5years
  time from randomization to death from any cause
disease-free survival (DFS) | 5 years
  The time between randomization and recurrence of disease or (for any reason) death.

CONTACTS AND LOCATIONS:
Locations (1):
- Chunling Jiang, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No